CLINICAL TRIAL: NCT03987048
Title: Cirrhotic Patients Admitted to the ICU With Septic Shock: Factors Predicting Short and Long-term Outcome
Brief Title: Cirrhotic Patients With Septic Shock
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: CSSM
Record Dates: First submitted 2019-05-03; First posted 2019-06-14 (Actual); Last update posted 2019-06-14 (Actual); Status verified 2019-05

CONDITIONS: Septic Shock; Cirrhosis
MeSH Terms: conditions — Shock, Septic; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cirrhotic patients with septic shock: All consecutive adult cirrhotic patients admitted to the ICU with septic shock from 2002 to 2013.
  Interventions: Other: Measure of short- and long-term mortality and analysis of independent predictors of short- and long-term mortality.

INTERVENTIONS:
Other: Measure of short- and long-term mortality and analysis of independent predictors of short- and long-term mortality. — Data were collected regarding medical background, medical condition and management, both at admission and during the ICU stay. These included demographics, clinical, biological and therapeutic data.
  Outcome at ICU discharge and at one year were also recorded.

SUMMARY:
Cirrhotic patients have a poor outcome in intensive care unit (ICU). Septic shock is a leading cause of ICU admission and death in this specific population. We performed a monocentric retrospective study; all cirrhotic patients admitted in the ICU with septic shock from 2002 to 2013 were included. The aim of the study was to identify prognostic factors for both short- and long-term mortality in these patients. Demographic, clinical and biological data, organ supports, and outcomes were collected. Univariate and multivariate analysis were carried out regarding both ICU and one-year mortality.

ELIGIBILITY:
Inclusion Criteria:

* age 18 or older
* diagnosis of cirrhosis
* diagnosis of septic shock at ICU admission

Exclusion Criteria:

* prior liver transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with cirrhosis who require ICU admission for septic shock
Sampling Method: Non-Probability Sample
Enrollment: 149 (Actual)
Dates: Start 2014-04 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Short-term outcome: analysis of independent predictors of ICU mortality rate. | Between ICU admission (from January 2002 to December 2013) and ICU discharge
  The predictors assessed independently are the clinical data, site of infection, biological data, liver scoring systems, organ failure, organ support and simplified acute physiology score (SAPS II), expressed in percentage of patients.
  The mortality rate is expressed in percentage of patients.
Long-term outcome: analysis of independent predictors of one-year mortality rate. | At one year after ICU admission (from January 2002 to December 2013)
  The predictors assessed independently are the independent predictors found to be related to the short-term mortality rate, expressed in percentage of patients.
  The mortality rate is expressed in percentage of patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Médecine Intensive-Réanimation, Hôpital Edouard Herriot (HCL), Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided